CLINICAL TRIAL: NCT07184385
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Two-arm Phase III Study to Assess the Efficacy of Human Umbilical Cord Blood (REGENECYTE) Infusion in Reducing Fatigue in Post-COVID Condition
Brief Title: A Study of Human Umbilical Cord Blood (REGENECYTE) Infusion in Patients With Post-COVID Condition
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: StemCyte, Inc. (Industry)
Responsible Party: Sponsor
Organization: StemCyte International, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCUS002
Record Dates: First submitted 2025-09-17; First posted 2025-09-19 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Long COVID; Post-COVID-19 Condition; Post-COVID Syndrome; Post-COVID Condition
Keywords: Post-COVID condition; Post-COVID syndrome; Long COVID; REGENECYTE; Post-COVID fatigue; Umbilical cord blood
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- REGENECYTE (Experimental): HPC, Cord Blood
  Interventions: Biological: REGENECYTE
- Placebo (Placebo Comparator): Normal Saline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: REGENECYTE — HPC, Cord Blood
  Arms: REGENECYTE
Biological: Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
REGENECYTE (HPC, Cord Blood) for treatment in patients with post-COVID.

DETAILED DESCRIPTION:
This is a two-arm, multi-center, double-blind, randomized, placebo-controlled phase III study. A total of 60 subjects with post-COVID will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18
* With post-COVID condition
* Has had a recent (within 7 days) negative SARS-CoV-2 test (an approved PCR or antigen test)
* Able to provide signed informed consent (by the subject or his/her legally authorized representative)
* Is willing and able to participate in all aspects of the study, including completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing a written informed consent

Exclusion Criteria:

* Neurological disorders prior to COVID-19 diagnosis
* With pre-existing terminal illness
* With known immune disease
* Is pregnant or breastfeeding
* Is currently participating in another investigational study or has been taking any other investigational product within the last 4 weeks before screening
* Has received any vaccination within 3 weeks prior to the first IP infusion or planning to receive vaccination during the treatment period
* Judged by the investigator to be not suitable for study participation, including but not limited to pre-existing chronic diseases
* Under the conditions that may increase risk of complications based on the medical judgment of the investigator and the parameters

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The change of efficacy | Week
  Change of efficacy evaluation

SECONDARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | Week
  Incidence of treatment-emergent adverse events (TEAEs)

IPD SHARING:
Plan to Share IPD: Undecided
All information supplied by StemCyte, Inc. in connection with this study and not previously published, is considered confidential information. This information includes, but is not limited to, the Investigator's Brochure, clinical protocol, case report forms and other scientific data. All data collected during the study are confidential. This confidential information shall remain the sole property of StemCyte, Inc. shall not be disclosed to others without the written consent of StemCyte, Inc. and shall not be used except in the performance of this study.